CLINICAL TRIAL: NCT06318169
Title: A Phase 3 Study to Evaluate the Efficacy and Safety of Pegozafermin in Subjects With Metabolic Dysfunction-Associated Steatohepatitis (MASH) and Fibrosis
Brief Title: A Study Evaluating the Efficacy and Safety of Pegozafermin in Participants With MASH and Fibrosis (ENLIGHTEN-Fibrosis)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: 89bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BIO89-100-131
Record Dates: First submitted 2024-03-13; First posted 2024-03-19 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Metabolic Dysfunction-Associated Steatotic Liver Disease (MASH) / Nonalcoholic Steatohepatitis (NASH) With Fibrosis
Keywords: Liver Diseases; Fatty Liver; Digestive System Diseases; Metabolic diseases; Metabolic Dysfunction-Associated Steatohepatitis; MASH; Steatohepatitis; Metabolic dysfunction-associated steatotic liver disease; MASLD; Nonalcoholic fatty liver disease; NAFLD; Fibrosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Diseases; Fatty Liver; Digestive System Diseases; Metabolic Diseases; Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pegozafermin Regimen 1 (Experimental)
  Interventions: Biological: Pegozafermin
- Pegozafermin Regimen 2 (Experimental)
  Interventions: Biological: Pegozafermin
- Placebo (Placebo Comparator): Matched Placebo will be administered in Regimens 1 and 2.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Pegozafermin — Subcutaneous injection
  Other Names: BIO89-100
  Arms: Pegozafermin Regimen 1; Pegozafermin Regimen 2
Other: Placebo — Subcutaneous injection
  Arms: Placebo

SUMMARY:
The study will assess the efficacy and safety of 2 dose regimens of pegozafermin compared to placebo for the treatment of liver fibrosis stage F2 or F3 in adult participants with MASH.

ELIGIBILITY:
Key Inclusion Criteria:

* Males or non-pregnant females aged between 18 and 80 years (inclusive) at time of signing the informed consent form (ICF)
* Biopsy-confirmed MASH with fibrosis stage F2 or F3
* Body mass index (BMI) at screening ≥25.0 kilograms (kg)/meters squared (m^2) (≥23 kg/m^2 for Asian participants).

Key Exclusion Criteria:

* Chronic liver diseases other than MASH
* Evidence of cirrhosis on screening liver biopsy
* Have type 1 diabetes or poorly controlled type 2 diabetes
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥250 units per liter (U/L)
* Participants taking vitamin E (>400 international units [IU]/day) or pioglitazone must be on stable dose for at least 6 months prior to Screening

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1350 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With at Least an Improvement of Fibrosis ≥1 Stage Without Worsening of Steatohepatitis at Week 52 | Week 52
  Worsening of steatohepatitis is defined as increase in non-alcoholic fatty liver disease (NAFLD) Activity Score (NAS) for ballooning, inflammation, or steatosis
Number of Participants With Resolution of Steatohepatitis Without Worsening of Fibrosis at Week 52 | Week 52
  Resolution of steatohepatitis is defined as total absence of ballooning (score=0) and absent or mild inflammation (score 0 to 1). Worsening of fibrosis is defined as progression of fibrosis by ≥1 stage.
Time to First Occurrence of Disease Progression | Up to 5 years
  Final analysis of the time to first occurrence of disease progression will be measured by a composite of protocol-specified clinical events

SECONDARY OUTCOMES:
Percent Change from Baseline in Alanine Aminotransferase at Week 52 | Baseline, Week 52
Absolute Change From Baseline in Enhanced Liver Fibrosis (ELF) Score at Week 52 | Baseline, Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Millie Gottwald, PharmD, Study Director — 89bio, Inc.
Locations (274):
- United States (114):
  - 89bio Clinical Study Site, Birmingham, Alabama
  - 89bio Clinical Study Site, Chandler, Arizona
  - 89bio Clinical Study Site, Flagstaff, Arizona
  - 89bio Clinical Study Site, Glendale, Arizona
  - 89bio Clinical Study Site, Tucson, Arizona
  - 89bio Clinical Study Site, Conway, Arkansas
  - 89bio Clinical Study Site, Little Rock, Arkansas
  - 89bio Clinical Study Site, North Little Rock, Arkansas
  - 89bio Clinical Study Site, Canoga Park, California
  - 89bio Clinical Study Site, Coronado, California
  - 89bio Clinical Study Site, Fountain Valley, California
  - 89bio Clinical Study Site, Fresno, California
  - 89bio Clinical Study Site, Gardena, California
  - 89bio Clinical Study Site, Huntington Park, California
  - 89bio Clinical Study Site, Inglewood, California
  - 89bio Clinical Study Site, La Jolla, California
  - 89bio Clinical Study Site, Lancaster, California
  - 89bio Clinical Study Site, Long Beach, California
  - 89bio Clinical Study Site, Los Angeles, California
  - 89bio Clinical Study Site, Montclair, California
  - 89bio Clinical Study Site, Orange, California
  - 89bio Clinical Study Site, Panorama City, California
  - 89bio Clinical Study Site, Pasadena, California
  - 89bio Clinical Study Site, Poway, California
  - 89bio Clinical Study Site, Rialto, California
  - 89bio Clinical Study Site, Santa Ana, California
  - 89bio Clinical Study Site, Stanford, California
  - 89bio Clinical Study Site, Victorville, California
  - 89bio Clinical Study Site, Colorado Springs, Colorado
  - 89bio Clinical Study Site, Littleton, Colorado
  - 89bio Clinical Study Site, Brandon, Florida
  - 89bio Clinical Study Site, Clermont, Florida
  - 89bio Clinical Study Site, Fort Myers, Florida
  - 89bio Clinical Study Site, Hialeah Gardens, Florida
  - 89bio Clinical Study Site, Jacksonville, Florida
  - 89bio Clinical Study Site, Jupiter, Florida
  - 89bio Clinical Study Site, Lady Lake, Florida
  - 89bio Clinical Study Site, Lakewood Rch, Florida
  - 89bio Clinical Study Site, Maitland, Florida
  - 89bio Clinical Study Site, New Port Richey, Florida
  - 89bio Clinical Study Site, Ocala, Florida
  - 89bio Clinical Study Site, Ocoee, Florida
  - 89bio Clinical Study Site, Sarasota, Florida
  - 89bio Clinical Study Site, Winter Park, Florida
  - 89bio Clinical Study Site, Athens, Georgia
  - 89bio Clinical Study Site, Dalton, Georgia
  - 89bio Clinical Study Site, Hammond, Indiana
  - 89bio Clinical Study Site, New Albany, Indiana
  - 89bio Clinical Study Site, South Bend, Indiana
  - 89bio Clinical Study Site, Iowa City, Iowa
  - 89bio Clinical Study Site, Topeka, Kansas
  - 89bio Clinical Study Site, Covington, Louisiana
  - 89bio Clinical Study Site, Houma, Louisiana
  - 89bio Clinical Study Site, Marrero, Louisiana
  - 89bio Clinical Study Site, New Orleans, Louisiana
  - 89bio Clinical Study Site, West Monroe, Louisiana
  - 89bio Clinical Study Site, Baltimore, Maryland
  - 89bio Clinical Study Site, Glen Burnie, Maryland
  - 89bio Clinical Study Site, Greenbelt, Maryland
  - 89bio Clinical Study Site, Burlington, Massachusetts
  - 89bio Clinical Study Site, Chesterfield, Michigan
  - 89bio Clinical Study Site, Wyoming, Michigan
  - 89bio Clinical Study Site, Ypsilanti, Michigan
  - 89bio Clinical Study Site, Rochester, Minnesota
  - 89bio Clinical Study Site, Flowood, Mississippi
  - 89bio Clinical Study Site, St Louis, Missouri
  - 89bio Clinical Study Site, Las Vegas, Nevada
  - 89bio Clinical Study Site, Florham Park, New Jersey
  - 89bio Clinical Study Site, Freehold, New Jersey
  - 89bio Clinical Study Site, Warren Township, New Jersey
  - 89bio Clinical Study Site, Albuquerque, New Mexico
  - 89bio Clinical Study Site, Carmel, New York
  - 89bio Clinical Study Site, New York, New York
  - 89bio Clinical Study Site, Charlotte, North Carolina
  - 89bio Clinical Study Site, Durham, North Carolina
  - 89bio Clinical Study Site, Fayetteville, North Carolina
  - 89bio Clinical Study Site, Morehead City, North Carolina
  - 89bio Clinical Study Site, Raleigh, North Carolina
  - 89bio Clinical Study Site, Winston-Salem, North Carolina
  - 89bio Clinical Study Site, Akron, Ohio
  - 89bio Clinical Study Site, Cleveland, Ohio
  - 89bio Clinical Study Site, Dayton, Ohio
  - 89bio Clinical Study Site, Liberty Township, Ohio
  - 89bio Clinical Study Site, Springboro, Ohio
  - 89bio Clinical Study Site, Westlake, Ohio
  - 89bio Clinical Study Site, East Greenwich, Rhode Island
  - 89bio Clinical Study Site, Charleston, South Carolina
  - 89bio Clinical Study Site, Columbia, South Carolina
  - 89bio Clinical Study Site, Chattanooga, Tennessee
  - 89bio Clinical Study Site, Cordova, Tennessee
  - 89bio Clinical Study Site, Hermitage, Tennessee
  - 89bio Clinical Study Site, Nashville, Tennessee
  - 89bio Clinical Study Site, Amarillo, Texas
  - 89bio Clinical Study Site, Austin, Texas
  - 89bio Clinical Study Site, Bellaire, Texas
  - 89bio Clinical Study Site, Brownsville, Texas
  - 89bio Clinical Study Site, Corpus Christi, Texas
  - 89bio Clinical Study Site, DeSoto, Texas
  - 89bio Clinical Study Site, Edinburg, Texas
  - 89bio Clinical Study Site, Farmers Branch, Texas
  - 89bio Clinical Study Site, Fort Sam Houston, Texas
  - 89bio Clinical Study Site, Fort Worth, Texas
  - 89bio Clinical Study Site, Garland, Texas
  - 89bio Clinical Study Site, Georgetown, Texas
  - 89bio Clinical Study Site, Houston, Texas
  - 89bio Clinical Study Site, Katy, Texas
  - 89bio Clinical Study Site, San Antonio, Texas
  - 89bio Clinical Study Site, Stafford, Texas
  - 89bio Clinical Study Site, Tomball, Texas
  - 89bio Clinical Study Site, Waco, Texas
  - 89bio Clinical Study Site, Ogden, Utah
  - 89bio Clinical Study Site, Richmond, Virginia
  - 89bio Clinical Study Site, Roanoke, Virginia
  - 89bio Clinical Study Site, Seattle, Washington
- Argentina (4):
  - 89bio Clinical Study Site, Buenos Aires
  - 89bio Clinical Study Site, Caba
  - 89bio Clinical Study Site, Capital Federal
  - 89bio Clinical Study Site, Pilar
- Australia (9):
  - 89bio Clinical Study Site, Brisbane, Queensland
  - 89bio Clinical Study Site, Herston, Queensland
  - 89bio Clinical Study Site, South Brisbane, Queensland
  - 89bio Clinical Study Site, Adelaide, South Australia
  - 89bio Clinical Study Site, Bedford Park, South Australia
  - 89bio Clinical Study Site, Clayton, Victoria
  - 89bio Clinical Study Site, Heidelberg, Victoria
  - 89bio Clinical Study Site, Perth, Western Australia
  - 89bio Clinical Study Site, Fitzroy
- Austria (5):
  - 89bio Clinical Study Site, Graz
  - 89bio Clinical Study Site, Innsbruck
  - 89bio Clinical Study Site, Klagenfurt
  - 89bio Clinical Study Site, Sankt Pölten
  - 89bio Clinical Study Site, Wels
- Belgium (5):
  - 89bio Clinical Study Site, Brussels
  - 89bio Clinical Study Site, Edegem
  - 89bio Clinical Study Site, Genk
  - 89bio Clinical Study Site, Ghent
  - 89bio Clinical Study Site, Jette
- Bulgaria (3):
  - 89bio Clinical Study Site, Gorna Oryahovitsa
  - 89bio Clinical Study Site, Sofia
  - 89bio Clinical Study Site, Stara Zagora
- Canada (7):
  - 89bio Clinical Study Site, Calgary, Alberta
  - 89bio Clinical Study Site, Vancouver, British Columbia
  - 89bio Clinical Study Site, Winnipeg, Manitoba
  - 89bio Clinical Study Site, London, Ontario
  - 89bio Clinical Study Site, Ottawa, Ontario
  - 89bio Clinical Study Site, Toronto, Ontario
  - 89bio Clinical Study Site, Vaughan, Ontario
- Czechia (3):
  - 89bio Clinical Study Site, Brno
  - 89bio Clinical Study Site, Ostrava
  - 89bio Clinical Study Site, Pilsen
- France (16):
  - 89bio Clinical Study Site, Amiens
  - 89bio Clinical Study Site, Angers
  - 89bio Clinical Study Site, Bordeaux
  - 89bio Clinical Study Site, Lille
  - 89bio Clinical Study Site, Limoges
  - 89bio Clinical Study Site, Lyon
  - 89bio Clinical Study Site, Montpellier
  - 89bio Clinical Study Site, Nantes
  - 89bio Clinical Study Site, Nice
  - 89bio Clinical Study Site, Paris
  - 89bio Clinical Study Site, Pierre-Bénite
  - 89bio Clinical Study Site, Strasbourg
  - 89bio Clinical Study Site, Toulouse
  - 89bio Clinical Study Site, Vandœuvre-lès-Nancy
  - 89bio Clinical Study Site, Vénissieux
  - 89bio Clinical Study Site, Villejuif
- Georgia (3):
  - 89bio Clinical Study Site, Batumi
  - 89bio Clinical Study Site, Tbilisi
  - 89bio_Clinical Study Site, Tbilisi
- Germany (6):
  - 89bio Clinical Study Site, Chemnitz
  - 89bio Clinical Study Site, Frankfurt am Main
  - 89bio Clinical Study Site, Freiburg im Breisgau
  - 89bio Clinical Study Site, Hanover
  - 89bio Clinical Study Site, Homburg
  - 89bio Clinical Study Site, Münster
- Hong Kong (2):
  - 89bio Clinical Study Site, Hong Kong
  - 89bio Clinical Study Site, Shatin
- India (6):
  - 89bio Clinical Study Site, Guwahati, Assam
  - 89bio Clinical Study Site, Kolkata, West Bengal
  - 89bio Clinical Study Site, Bhubaneswar
  - 89bio Clinical Study Site, Gujrāt
  - 89bio Clinical Study Site, Nagpur
  - 89bio Clinical Study Site, Wardha
- Israel (8):
  - 89bio Clinical Study Site, Afula
  - 89bio Clinical Study Site, Beersheba
  - 89bio Clinical Study Site, Haifa
  - 89bio Clinical Study Site, Jerusalem
  - 89bio Clinical Study Site, Nahariya
  - 89bio Clinical Study Site, Petah Tikva
  - 89bio Clinical Study Site, Ramat Gan
  - 89bio Clinical Study Site, Tel Aviv
- Italy (9):
  - 89bio Clinical Study Site, Bergamo
  - 89bio Clinical Study Site, Milan
  - 89bio Clinical Study Site, Modena
  - 89bio Clinical Study Site, Napoli
  - 89bio Clinical Study Site, Novara
  - 89bio Clinical Study Site, Palermo
  - 89bio Clinical Study Site, Roma
  - 89bio Clinical Study Site, Rome
  - 89bio Clinical Study Site, Torino
- Japan (14):
  - 89bio Clinical Study Site, Maebashi, Gunma
  - 89bio Clinical Study Site, Sapporo, Hokkaido
  - 89bio Clinical Study Site, Hizume, Iwate
  - 89bio Clinical Study Site, Kawasaki, Kanagawa
  - 89bio Clinical Study Site, Yokohama, Kanagawa
  - 89bio Clinical Study Site, Ehime
  - 89bio Clinical Study Site, Fukuoka
  - 89bio Clinical Study Site, Gifu
  - 89bio Clinical Study Site, Kumamoto
  - 89bio Clinical Study Site, Nagano
  - 89bio Clinical Study Site, Okayama
  - 89bio Clinical Study Site, Osaka
  - 89bio Clinical Study Site, Saga
  - 89bio Clinical Study Site, Sapporo
- Mexico (7):
  - 89bio Clinical Study Site, Chihuahua City
  - 89bio Clinical Study Site, Cuautitlán Izcalli
  - 89bio Clinical Study Site, Jalisco
  - 89bio Clinical Study Site, Mexico City
  - 89bio Clinical Study Site, Morelos
  - 89bio Clinical Study Site, Nuevo León
  - 89bio Clinical Study Site, Yucatán
- Netherlands (3):
  - 89bio Clinical Study Site, Rotterdam, South Holland
  - 89bio Clinical Study Site, Amsterdam
  - 89bio Clinical Study Site, Utrecht
- Poland (6):
  - 89bio Clinical Study Site, Katowice
  - 89bio Clinical Study Site, Krakow
  - 89bio Clinical Study Site, Lodz
  - 89bio Clinical Study Site, Mysłowice
  - 89bio Clinical Study Site, Warsaw
  - 89bio Clinical Study Site, Wroclaw
- Puerto Rico (2):
  - 89bio Clinical Study Site, Mayagüez
  - 89bio Clinical Study Site, San Juan
- 89bio Clinical Study Site, Singapore, Singapore
- South Africa (3):
  - 89bio Clinical Study Site, Cape Town
  - 89bio Clinical Study Site, Johannesburg
  - 89bio Clinical Study Site, Worcester
- South Korea (5):
  - 89bio Clinical Study Site, Busan
  - 89bio Clinical Study Site, Daegu
  - 89bio Clinical Study Site, Gyeonggi-do
  - 89bio Clinical Study Site, Incheon
  - 89bio Clinical Study Site, Seoul
- Spain (9):
  - 89bio Clinical Study Site, Barcelona
  - 89bio Clinical Study Site, Córdoba
  - 89bio Clinical Study Site, Madrid
  - 89bio Clinical Study Site, Majadahonda
  - 89bio Clinical Study Site, Málaga
  - 89bio Clinical Study Site, Pontevedra
  - 89bio Clinical Study Site, Santander
  - 89bio Clinical Study Site, Santiago de Compostela
  - 89bio Clinical Study Site, Seville
- Taiwan (3):
  - 89bio Clinical Study Site, Chiayi City
  - 89bio Clinical Study Site, Kaohsiung City
  - 89bio Clinical Study Site, Taipei
- Turkey (Türkiye) (8):
  - 89bio Clinical Study Site, Adana
  - 89bio Clinical Study Site, Ankara
  - 89bio Clinical Study Site, Bursa
  - 89bio Clinical Study Site, Fatih
  - 89bio Clinical Study Site, Istanbul
  - 89bio Clinical Study Site, Merkez
  - 89bio Clinical Study Site, Sarıçam
  - 89bio Clinical Study Site, Umraniye
- United Kingdom (13):
  - 89bio Clinical Study Site, High Wycombe, Buckinghamshire
  - 89bio Clinical Study Site, Bristol
  - 89bio Clinical Study Site, Glasgow
  - 89bio Clinical Study Site, Hull
  - 89bio Clinical Study Site, London
  - 89bio Clinical Study Site, Oxford
  - 89bio Clinical Study Site, Portsmouth
  - 89bio Clinical Study Site, Preston
  - 89bio Clinical Study Site, Southampton
  - 89bio Clinical Study Site, Stockton
  - 89bio Clinical Study Site, Sunderland
  - 89bio Clinical Study Site, Swansea
  - 89bio Clinical Study Site, York